CLINICAL TRIAL: NCT02046694
Title: A Pilot Study of Allopurinol As A Modifier of 6-MP Metabolism in Pediatric ALL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1357; J1357 (Other: SKCCC at Johns Hopkins); NA_00084984 (Other: JHMIRB)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: acute lymphoblastic leukemia; ALL; pediatric; maintenance; allopurinol; 6-MP; 6-mercaptopurine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allopurinol (Experimental): Patients will stop taking their 6-MP and methotrexate at week 0. One week later (week 1), patients will begin allopurinol daily (100 mg for weight >30 kg, 50 mg for weight ≤30 kg) and will restart 6-MP and methotrexate at 50 percent of the most recent dose. Patients will continue taking allopurinol in combination with 6-MP and methotrexate for the duration of the study (total of 8 weeks). Dose adjustments of 6-MP and methotrexate will be directed by the guidelines outlined in the study protocol.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — At week 1, patients will begin allopurinol daily (100 mg for weight >30 kg, 50 mg for weight ≤30 kg) and will restart 6-MP and methotrexate at 50 percent of the most recent dose. Patients will continue taking allopurinol in combination with 6-MP and methotrexate for the duration of the study (total of 8 weeks).
  Other Names: Zyloprim

SUMMARY:
This research is being done to determine if allopurinol can change the metabolism of the oral chemotherapeutic medication 6-mercaptopurine (6-MP) in children with acute lymphoblastic leukemia (ALL). 6-MP is originally started at a standard dose in children with ALL, but the dose is adjusted according to the absolute neutrophil count (ANC). Occasionally, 6-MP doses need to be increased in order to get the ANC into a specific target range. Also, increasing the 6-MP dose can lead to unwanted side effects, such as inflammation of the liver as shown by increases in laboratory values (ALT, aspartate aminotransferase (AST), bilirubin), nausea, and abdominal discomfort. Previous studies in children with inflammatory bowel disease has shown that combining allopurinol with 6-MP can decrease side effects associated with high doses of 6-MP and also increase the efficacy of 6-MP. Allopurinol is approved by the Food and Drug Administration for the treatment of tumor lysis syndrome in ALL. Through this research study, the investigators hope to show that the combination of allopurinol and 6-MP will be safe, tolerable, and effective in children with ALL.

DETAILED DESCRIPTION:
* Patients will have several visits to the Pediatric Oncology outpatient clinic. Each visit will consist of a physical examination and laboratory evaluation. Each laboratory evaluation will consist of taking approximately 10-15 milliliters of blood (or approximately three teaspoons). These clinic visits may actually coincide with clinic visits that were previously scheduled according to the patient's treatment protocol.
* At the first study visit, patients will have a physical examination and laboratory evaluation. At that visit, patients will be asked to stop taking 6-MP and methotrexate.
* At the second study visit, which is one week later, patients will again have a physical examination and laboratory evaluation. The investigators will prescribe allopurinol and restart 6-MP and methotrexate at half of the patient's previous doses.
* Clinic visits for physical examination and laboratory evaluation will be scheduled every 1-2 weeks for a total of 5 more visits. Doses of allopurinol, 6-MP, and methotrexate may be adjusted at these visits based on laboratory values or clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated in the maintenance phase of therapy for pediatric ALL
* Age ≤30 years
* 6-MMP:6-TGN ratio ≥40 within 21 days prior to enrollment
* 6-MMP ≥12,000/8x108 red blood cells (RBC) within 21 days prior to enrollment
* One of the following within 21 days prior to enrollment:

  1. ANC persistently ≥1500/mm3 (as measured by 3 CBCs done over 6 weeks or 2 successive monthly complete blood counts (CBCs) despite 6-MP ≥150% of Children's oncology group (COG) dosing OR
  2. Evidence of ≥ Grade 3 hepatotoxicity with one of the following:

     ALT ≥5x upper limit of normal (based on institutional standards) AST ≥5x upper limit of normal (based on institutional standards) Direct bilirubin ≥5x upper limit of normal (based on institutional standards) OR
  3. Evidence of ≥ Grade 2 gastrointestinal toxicity (including, but not limited to: nausea, vomiting, anorexia, gastrointestinal pain)

Exclusion Criteria:

* Allergy to allopurinol
* Active relapse of ALL or lymphoblastic lymphoma
* Currently enrolled on any therapeutic research study for the treatment of ALL or lymphoblastic lymphoma
* Known history of chronic liver disease (other than Gilbert's syndrome)
* Pregnant or breastfeeding females

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Absolute neutrophil count | 8 weeks
  Absolute neutrophil count (ANC) measured 8 weeks after the addition of allopurinol (study week 9).

SECONDARY OUTCOMES:
Feasibility of the addition of allopurinol to ALL maintenance therapy | 8 weeks
  Allopurinol compliance rate during ALL maintenance therapy.
Safety of the addition of allopurinol to ALL maintenance therapy | 8 weeks
  Occurence of grade 4 adverse events that are possibly, probably, or definitely attributable to allopurinol.
Effects of allopurinol on liver function tests | 8 weeks
  Measurement of ALT, AST, and direct bilirubin before and after adding allopurinol.
Alteration of 6-MP metabolism through the addition of allopurinol | 8 weeks
  Measurement of 6-thioguanine (6-TGN) and 6-methylmercaptopurine (6-MMP) before and after adding allopurinol.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Cooper, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Pui CH, Evans WE. Treatment of acute lymphoblastic leukemia. N Engl J Med. 2006 Jan 12;354(2):166-78. doi: 10.1056/NEJMra052603. No abstract available. PMID 16407512
- [Background] Ansari A, Elliott T, Baburajan B, Mayhead P, O'Donohue J, Chocair P, Sanderson J, Duley J. Long-term outcome of using allopurinol co-therapy as a strategy for overcoming thiopurine hepatotoxicity in treating inflammatory bowel disease. Aliment Pharmacol Ther. 2008 Sep 15;28(6):734-41. doi: 10.1111/j.1365-2036.2008.03782.x. PMID 19145729
- [Background] Rahhal RM, Bishop WP. Initial clinical experience with allopurinol-thiopurine combination therapy in pediatric inflammatory bowel disease. Inflamm Bowel Dis. 2008 Dec;14(12):1678-82. doi: 10.1002/ibd.20522. PMID 18521913
- [Background] Sparrow MP, Hande SA, Friedman S, Lim WC, Reddy SI, Cao D, Hanauer SB. Allopurinol safely and effectively optimizes tioguanine metabolites in inflammatory bowel disease patients not responding to azathioprine and mercaptopurine. Aliment Pharmacol Ther. 2005 Sep 1;22(5):441-6. doi: 10.1111/j.1365-2036.2005.02583.x. PMID 16128682
- [Background] Sparrow MP, Hande SA, Friedman S, Cao D, Hanauer SB. Effect of allopurinol on clinical outcomes in inflammatory bowel disease nonresponders to azathioprine or 6-mercaptopurine. Clin Gastroenterol Hepatol. 2007 Feb;5(2):209-14. doi: 10.1016/j.cgh.2006.11.020. PMID 17296529
- [Background] Koren G, Ferrazini G, Sulh H, Langevin AM, Kapelushnik J, Klein J, Giesbrecht E, Soldin S, Greenberg M. Systemic exposure to mercaptopurine as a prognostic factor in acute lymphocytic leukemia in children. N Engl J Med. 1990 Jul 5;323(1):17-21. doi: 10.1056/NEJM199007053230104. PMID 2355954
- [Background] Balis FM, Holcenberg JS, Poplack DG, Ge J, Sather HN, Murphy RF, Ames MM, Waskerwitz MJ, Tubergen DG, Zimm S, Gilchrist GS, Bleyer WA. Pharmacokinetics and pharmacodynamics of oral methotrexate and mercaptopurine in children with lower risk acute lymphoblastic leukemia: a joint children's cancer group and pediatric oncology branch study. Blood. 1998 Nov 15;92(10):3569-77. PMID 9808549
- [Background] Pui CH, Mullighan CG, Evans WE, Relling MV. Pediatric acute lymphoblastic leukemia: where are we going and how do we get there? Blood. 2012 Aug 9;120(6):1165-74. doi: 10.1182/blood-2012-05-378943. Epub 2012 Jun 22. PMID 22730540
- [Background] Zimm S, Collins JM, O'Neill D, Chabner BA, Poplack DG. Inhibition of first-pass metabolism in cancer chemotherapy: interaction of 6-mercaptopurine and allopurinol. Clin Pharmacol Ther. 1983 Dec;34(6):810-7. doi: 10.1038/clpt.1983.254. PMID 6580097
- [Background] Elion GB. The purine path to chemotherapy. Science. 1989 Apr 7;244(4900):41-7. doi: 10.1126/science.2649979.
- [Background] Brackett J, Schafer ES, Leung DH, Bernhardt MB. Use of allopurinol in children with acute lymphoblastic leukemia to reduce skewed thiopurine metabolism. Pediatr Blood Cancer. 2014 Jun;61(6):1114-7. doi: 10.1002/pbc.24913. Epub 2013 Dec 27. PMID 24376133
- [Background] Jharap B, Seinen ML, de Boer NK, van Ginkel JR, Linskens RK, Kneppelhout JC, Mulder CJ, van Bodegraven AA. Thiopurine therapy in inflammatory bowel disease patients: analyses of two 8-year intercept cohorts. Inflamm Bowel Dis. 2010 Sep;16(9):1541-9. doi: 10.1002/ibd.21221. PMID 20155846